CLINICAL TRIAL: NCT00621907
Title: Levobupivacïne Into Post-analgesia : Randomized Monocentric Study Against Placebo
Brief Title: Study : LEVOBUPIVACAINE Versus Placebo
Acronym: LEVOBU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Clément CAILLAUX, Centre Hospitalo-Universitaire de Saint-Etienne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0708097; 2007-006275-36
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Pain
Keywords: randomized; analgesic; caesarean scars; locoregional anaesthesia; infiltration; levobupivacaïne; Chirocaïne; caesarian; unique administration; post-caesarian analgesic
MeSH Terms: conditions — Pain | interventions — Levobupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): patient who received levobupivacaïne
  Interventions: Drug: chirocaine (Levobupivacaine)
- 2 (Placebo Comparator): patient who received placebo
  Interventions: Drug: sodium chloride

INTERVENTIONS:
Drug: chirocaine (Levobupivacaine) — levobupivacaine 0,5 % 30 ml infiltration (150 mg)
  Arms: 1
Drug: sodium chloride — sodium chloride : 0,9% 30 ml
  Arms: 2

SUMMARY:
The locoregional anaesthesia is increasingly important in surgical practice, often allowing to simplify per- and post-operative analgesia. caesarian occurs in 20 % of delivery leading to a longer hospitalization because of the pain resulting from the surgery. The Levobupivacaïne (Chirocaïne) administered through catheters placed in the caesarean scars, showed its efficiency in post-operative analgesia.

Method : realization of a double blind prospective randomized study, control versus placebo Purpose : to show that the local administration of a unique dose of analgesia reduce the post-operative pain with a little or non-invasive technique

DETAILED DESCRIPTION:
The study will be done at the department of Obstétric and gynecology, in the CHU of Saint-Etienne. It will include all patients requiring a caesarean without any contraindication.

All the patients requiring a urgent or a very urgent caesarean will be excluded because a rapid consent can't be obtained and the product preparation can't be done.

Inclusion after information and minimum one hour of time for consideration. Randomization : the teatment group will be randomized according to the patient number : control versus placebo : 70 patients in the group infiltration of levobupivacaïne and 70 patients in the group infiltration of a placebo. Every product will be prepared in a 30 ml syringe filled with levobupivacaïne or 0,9 % sodium chloride depending on the group of randomization. All patients will get their caesarean according to the same technique, then, before the cutaneous close, the product will be injected in the caesarean wall.

Fllow-up : supervision of the pain (morphine consumption, VAS) and of undesirable effects.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* all patients requiring a non-urgent caesarian done according to the Misgav-Ladach technique

Exclusion Criteria:

* Patients requiring very urgent caesarian
* allergic to levobupivacaïne
* with previous history of alcoholism or drug addiction
* with severe hypotension or an ischemic cardiopathy badly compensated or thyrotoxicoses
* treated with first generation of IMAO (monoamine oxidase inhibitor) or with anti-arrhytmia drugs with anesthesic activity

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2008-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
analgesic consumption of level 3 in the two treated groups | 24 hours

SECONDARY OUTCOMES:
visual analogic scale (VAS) at rest or on rising, early rehabilitation, residual pain 2 months after the operation | hours : 1, 2, 3, 4, 5, 6, 8, 12, 24, 48 and at 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Céline CHAULEUR, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- University Hospital, Saint-Etienne, France

REFERENCES:
- [Derived] Corsini T, Cuvillon P, Forgeot A, Chapelle C, Seffert P, Chauleur C. [Single-dose intraincisional levobupivacaine infiltration in caesarean postoperative analgesia: a placebo-controlled double-blind randomized trial]. Ann Fr Anesth Reanim. 2013 Jan;32(1):25-30. doi: 10.1016/j.annfar.2012.10.035. Epub 2012 Dec 21. French. PMID 23260628